CLINICAL TRIAL: NCT06414382
Title: Pilot Study on Koebner Induction in Patients With Plaque Psoriasis
Brief Title: PSODEEP2 Pilot Study on Koebner Induction in Psoriasis
Acronym: PSODEEP2PIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: University of Copenhagen (Other); Lund University (Other)
Responsible Party: Principal Investigator, Albert Duvetorp, Principal Investigator, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSODEEP2PIL
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis Vulgaris; Koebner Phenomenon

STUDY DESIGN:
Intervention Model Description: Koebner phenomena will be induced using tape-stripping or tape-stripping and micro needling. Koebner development will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Koebner induction (Experimental): Koebner will be induced on area 22mm in diameter on upper bilateral arms and anterior bilateral thighs.
  Interventions: Other: Tape-stripping

INTERVENTIONS:
Other: Tape-stripping — 22mm tapes x 40 will be attached and removed to skin of all for limbs (tape stripping). On left arm and leg skin will also be subject to micro needling.
  Other Names: Micro-needling

SUMMARY:
Patients (n=15) with skin psoriasis, minimum age 18 years, without systemic immunomodulatory treatment will be subject to Koebner induction on arms and legs given that they have given written consent and that they have self-reported Koebner.

DETAILED DESCRIPTION:
PSODEEP2 PILOT STUDY

Study subject recruitation:

Individuals fulfilling inclusion and exclusion criteria will be identified and contacted from the PSODEEP1 study (ethical application2023-00571-02 and 2022-02835-01), advert in social media, advert in newsletter/magazine sent out by patients organizations (Ung med Psoriasis or Psoriasisförbundet) or through direct contact with patients visits in dermatology department (n = 15).

Inclusion criteria:

Psoriasis skin disease. Self-reported experience of Koebner phenomena. Age 18 years or older. Ability to comprehend study information. Signed and dated informed consent.

Exclusion criteria:

Ongoing or planned systemic immunomodulatory treatment. Ongoing or planned narrowband UVB or PUVA treatment. Lack of suitable non-lesional skin on proximal arm or thigh due to extensive psoriatic disease.

Intervention:

Non-lesional skin 22mm in diameter on proximal arm or thigh at least 5 cm from the closest psoriasis lesion will be identified and marked bilaterally using a surgical skin marker. The skin sites will be documented using digital photography and the photos will be stored in REDCap (project-redcap.org). Tape will be attached and removed from the skin 40 times at all 4 sites using D-squame 22mm sampling discs and D-squame pressure applicator. Tapes are to be removed using tweezers by research staff wearing nitrile/vinyl gloves and moved to D- squame Disc Carrier which are coded/labelled so that each sampling disc has a unique code. The codes are transferred to REDCap together with study subjects background information. Tapes are transferred to -70 storage in labelled cryotubes (stored one disc per tube) prior to proteomic analysis. Taped stripped skin on left arm and left thigh is then stimulated with microneedle device (Dermapen 4) set at 0,8 mm. Study subjects are asked to contact the research group if or when psoriasis develop at any of the four stimulated sites. Study subjects will be instructed to inspect skin once daily at a minimum. If uncertainty arises as to whether psoriasis has developed it will be possible to book an appointment for skin evaluation. If psoriasis develops a second appointment will be booked. At the second appointment all 4 locations will be documented using digital photography (and stored in REDCap). Locations will be re-sampled using 10 D- squame 22mm sampling discs per location. At locations showing signs of psoriasis development, induration, erythema and scaling will be assessed and recorded in REDCap (0- 4 points). In local anesthesia, a 4mm punch biopsy will be performed from developed psoriasis lesions (K+) (Koebner positive) and put in Eppendorf tube before being frozen on dry ice, labelled with unique code and transferred to - 70 freezer before further analysis. If no psoriasis develops then the study subjects will be booked for appointment 2 approximately day 21 after Koebner induction. For these subjects stratum corneum skin sampling will be performed at all four sites using 10 D-squame 2mm sampling discs transferred to D-squame Disc Carrier and then to cryotubes for storage at - 70 °C.

Bioanalysis:

For proteomic analysis, proteins will be lysed directly on the tape strips and prepared according to previously described protocol after which liquid chromatography-mass spectrometry will be performed (21).

Punch biopsies from developing or early psoriasis lesions will be analyzed accordingly to validate psoriasis development including histological assessment of signs of psoriasis (parakeratosis, psoriasiform hyperplasia, epidermal neutrophilic infiltration, dilated vessels in papillary dermis, loss of stratum granulosum). Additionally modern techniques analyzing the transcriptome, proteome and epigenome will be used to assess psoriasis development.

Study significance:

The PILOT study aims to answer research questions:

* Will the addition of micro-needling to tape-stripping increase Koebner reactivity in non-lesional psoriasis skin?
* Does Koebner-reactivity differ between proximal arm and proximal leg?

The answer to these questions are essential to determine the optimal intervention of the main study. The method and location that results in the higher proportion of Koebner positive reactions will be selected for the main study. It will also provide preliminary proteomic data which can facilitate a more accurate sample size calculation for main study.

ELIGIBILITY:
Inclusion Criteria:

* Self reported Koebner
* Diagnosis of skin psoriasis

Exclusion Criteria:

* Systemic immunomodulatory treatment (including narrowband UVB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-07 (Estimated); Primary Completion 2024-12-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Positive Koebner Phenomena (K+) | 7-21 days after induction
  Psoriasis lesion develops at site of provocation/induction
Negative Koebner Phenomena (K-) | 21 days after induction
  No psoriasis lesion develops at site of provocation/induction

SECONDARY OUTCOMES:
Stratum corneum proteomics | At baseline and at time of K+ assessment or day 21 if K-
  Mass spectrometry of stratum corneum at koebner induction sites

CONTACTS AND LOCATIONS:
Overall Officials: Liv Eidsmo, Professor, Study Director — Copenhagen University SIC, Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
This is a pilot study necessary for selection of suitable method in subsequent follow up study. Data sharing outside research group has not been part of the ethical approval´s description of data handling. These two reasons are behind the "no".